CLINICAL TRIAL: NCT01030315
Title: A Randomized, Double-Blind, Placebo-Controlled, Sequential Dose Escalation Study of the Safety, Pharmacodynamics and Pharmacokinetics of Single Intravenous Doses of HM10760A in Healthy Adult Caucasian and Japanese Subjects
Brief Title: A Study of HM10760A (Long-acting Erythropoietin) in Healthy Adult Caucasian and Japanese Subjects
Acronym: EPO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-HM10760A-101
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: Erythropoietin; Long-acting; EPO

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): The lowest dose level of HM10760A
  Interventions: Drug: HM10760A or placebo
- Cohort 2 (Experimental): Second dose level of HM10760A
  Interventions: Drug: HM10760A or placebo
- Cohort 3 (Experimental): Third dose level of HM10760A
  Interventions: Drug: HM10760A or placebo
- Cohort 4 (Experimental): Fourth dose level of HM10760A
  Interventions: Drug: HM10760A or placebo
- Cohort 5 (Experimental): The highest dose level of HM10760A
  Interventions: Drug: HM10760A or placebo

INTERVENTIONS:
Drug: HM10760A or placebo — Once, 0.04 mcg/kg to 2.0mcg/kg once intravenously

SUMMARY:
Study design:

* Phase I, first-in-human, randomized, double-blind, placebo-controlled, sequential dose escalation study of intravenously administered HM10760A in healthy adult Caucasian and Japanese subjects. Up to 5 dose level cohorts are planned. In each dose level cohort, subjects will be randomized to receive a single dose of HM10760A or placebo.

Primary Objective:

* To evaluate safety profile of single intravenous (IV) dose levels of HM10760A in healthy adult Caucasian and Japanese subjects.

DETAILED DESCRIPTION:
Secondary Objectives:

* To evaluate the dose response relationship of a single IV dose of HM10760A on pharmacodynamic parameters
* To assess the immunogenicity of a single IV dose of HM10760A.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian and Japanese male and/or female volunteers
* Age 18 to 55 years
* Hemoglobin of >12 g/dL and <16 g/dL for male subjects, >10 g/dL and <14 g/dL for female Caucasian subjects

Exclusion Criteria:

* Prior exposure to EPO, darbepoetin, other EPO support proteins
* hypersensitivity to EPO, darbepoetin, E.coli derived proteins
* Hemoglobinopathy
* SBP > 140 mmHg or < 90 mmHg or DBP > 95 mmHg
* Chronic, uncontrolled, or symptomatic inflammatory disease
* Malignancy(except non-melanoma skin cancer)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety data, including physical examinations, laboratory evaluation, ECGs, vital signs, adverse events, and endogenous erythropoietin level. | 84 days after the investigational drug administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanmi Clinical, US, California, United States